CLINICAL TRIAL: NCT02685033
Title: A Phase 2, Single-center, Open-label, Randomized, Comparator-controlled Trial of the Safety and Efficacy of Dalbavancin Versus Active Comparator in Adult Patients With Osteomyelitis Known or Suspected to be Due to Gram-Positive Organisms
Brief Title: Study on the Safety and Efficacy of Dalbavancin Versus Active Comparator in Adult Participants With Osteomyelitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durata Therapeutics Inc., an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAL-MD-04
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Osteomyelitis
Keywords: Osteomyelitis; dalbavancin; antibiotic
MeSH Terms: conditions — Osteomyelitis | interventions — dalbavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dalbavancin (Experimental): Dalbavancin 1500 mg, intravenous (IV) administration over 30 minutes on Day 1 and Day 8. If creatinine clearance was < 30 milliliters per minute (mL/min) and participant was not receiving regular hemodialysis or peritoneal dialysis, dalbavancin dose was decreased to 1000 mg.
  Interventions: Drug: Dalbavancin
- Standard of Care (Active Comparator): Antibiotic consistent with Standard of Care (SOC), based on baseline pathogen, for 4 to 6 weeks.
  Interventions: Drug: Comparator

INTERVENTIONS:
Drug: Dalbavancin
  Other Names: Dalvance®; Xydalba™
  Arms: Dalbavancin
Drug: Comparator
  Arms: Standard of Care

SUMMARY:
This clinical study will be a single-center, randomized, open-label, active-controlled, parallel-group study comparing dalbavancin to standard of care (SOC) therapy in osteomyelitis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of osteomyelitis (first episode) defined by:
* Pain or point tenderness upon palpation or probing to bone
* Plain radiograph or Magnetic resonance imaging (MRI) consistent with osteomyelitis (indistinctly marginated edema-like pattern of bone marrow hypointensity on unenhanced T1-weighted sequences, hyperintensity on fat-saturated T2-weighted and Short tau inversion recovery (STIR) sequences and/or abnormal enhancement on gadolinium-enhanced fat-saturated T2-weighted sequences, with or without visible periostitis or cortical bone destruction) OR Gram-positive cocci documented on a baseline Gram-stain from a bone specimen
* Elevated C-reactive protein (CRP) (low sensitivity) above the upper limit of normal (ULN) (reference range for low sensitivity CRP is 3-10 mg/L)
* Participants must be willing and able, if discharged from the hospital, to return to the hospital or a designated clinic for scheduled visits, treatment, laboratory tests, and other outpatient procedures as required by the protocol.

Exclusion Criteria:

* Treatment with an investigational drug within 30 days preceding the first dose of investigational product.
* Receipt of > 24 hours of potentially effective IV antibacterial therapy for osteomyelitis within 96 hours of randomization, unless the pathogen isolated was documented to be Methicillin-resistant Staphylococcus aureus (MRSA) that was resistant to the administered antibiotic.
* A prior episode of osteomyelitis, or a failed course of therapy for osteomyelitis.
* Infection associated with a burn wound, with a sacral decubitus ulcer, or with multiple sites of osteomyelitis.
* Septic arthritis that is non-contiguous to osteomyelitis, as diagnosed by isolation of a pathogen from synovial fluid culture.
* Immunosuppression/immune deficiency
* Evidence of Gram-negative bacteria by Gram stain in the absence of Gram-positive organisms.
* Gram-negative bacteremia
* Patients with concomitant endocarditis, necrotizing fasciitis, or prosthetic material at the site of infection at the time of study initiation.
* Infection due to an organism known prior to study entry to not be susceptible to dalbavancin (dalbavancin mean inhibitory concentration [MIC] > 0.12 μg/mL) or vancomycin (vancomycin MIC > 2 μg/mL).
* Concomitant systemic antibacterial therapy for Gram-positive infections (eg, rifampin, gentamicin).
* Known or suspected hypersensitivity to glycopeptide antibiotics.
* Patients with a rapidly fatal illness, who are not expected to survive for 3 months.
* Pregnant or nursing females; positive urine (or serum) pregnancy test at Screening (pre-menopausal females only) or after admission (prior to dosing)
* Sexually active females of childbearing potential who are unwilling or unable to use an acceptable method of contraception from at least the first dose of study drug until the last pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Urania Rappo, MD, MS, PharmD, Study Director — Allergan
Locations (1):
- Allergan Investigative Site 001, Cherkasy, Ukraine

REFERENCES:
- [Derived] Rappo U, Puttagunta S, Shevchenko V, Shevchenko A, Jandourek A, Gonzalez PL, Suen A, Mas Casullo V, Melnick D, Miceli R, Kovacevic M, De Bock G, Dunne MW. Dalbavancin for the Treatment of Osteomyelitis in Adult Patients: A Randomized Clinical Trial of Efficacy and Safety. Open Forum Infect Dis. 2018 Dec 10;6(1):ofy331. doi: 10.1093/ofid/ofy331. eCollection 2019 Jan. PMID 30648126

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalbavancin | Standard of Care
Started | 70 | 10
Completed | 67 | 8
Not Completed | 3 | 2
Not completed — Withdrawal of Consent | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all intent-to-treat (ITT) participants who received any amount of randomized medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalbavancin | Standard of Care | Total
Number analyzed (Participants) | 70 | 10 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (13.3) | 54.4 (15.3) | 49.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 59 | 5 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 70 | 10 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 70 | 10 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response at Day 42 in the Clinically Evaluable (CE) Population
Description: Clinical response was either cure, failure or indeterminate. A cure was defined as recovery without need for additional antibiotic therapy. A failure was defined as the requirement of additional antibiotic therapy for no response or worsening after improvement, new purulence, amputation due to progression of infection (from initiation of study drug to outcome assessment visit), requiring >6 weeks of antibiotic therapy for participants in the standard of care arm or death (for any reason). Indeterminate was defined as lost to follow-up or amputation due to vascular insufficiency (from initiation of study drug to outcome assessment visit).
Time Frame: Day 42
Population: CE-D42 population included all modified intent-to-treat (mITT) participants who met specific conditions for evaluability at Day 42 (D42).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 67 | 8
percentage of participants
  Clinical Cure | 97.0 [89.6 to 99.6] | 87.5 [47.3 to 99.7]
  Clinical Failure | 0.0 [NA to NA] — As per protocol, 95% Confidence Interval (CI) was only calculated for outcome of clinical cure. | 12.5 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.
  Indeterminate | 3.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 0.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.

2. Secondary Outcome: Percentage of Participants With Clinical Improvement at Day 21 in the mITT Population
Description: Clinical improvement was defined as no worsening of pain from baseline, if present (subjective pain and/or point tenderness), and improvement in inflammation (as measured by C-reactive protein [CRP]).
Time Frame: Baseline to Day 21
Population: mITT population included all ITT participants who received any amount of randomized medication and met the criteria for known or suspected Gram-positive osteomyelitis. Participants from whom only a Gram-negative pathogen was isolated from blood and/or bone culture were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 67 | 8
percentage of participants | 94.0 [85.4 to 98.3] | 62.5 [24.5 to 91.5]

3. Secondary Outcome: Percentage of Participants With Clinical Improvement at Day 21 in the CE Population
Description: as for outcome 2
Time Frame: Baseline to Day 21
Population: CE-D21 population included all mITT (modified intent-to-treat) participants who met specific conditions for evaluability at Day 21 (D21).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 67 | 8
percentage of participants | 94.0 [85.4 to 98.3] | 62.5 [24.5 to 91.5]

4. Secondary Outcome: Percentage of Participants With Clinical Response at Day 42 in the mITT Population
Description: as for outcome 1
Time Frame: Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 67 | 8
percentage of participants
  Clinical Cure | 97.0 [89.6 to 99.6] | 87.5 [47.3 to 99.7]
  Clinical Failure | 0.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 12.5 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.
  Indeterminate | 3.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 0.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.

5. Secondary Outcome: Percentage of Participants With Clinical Response at Day 42 in the Microbiological Modified Intent-to-Treat (Micro-mITT) Population
Description: as for outcome 1
Time Frame: Day 42
Population: Micro-mITT population included mITT participants with a Gram-positive pathogen isolated from blood and/or bone specimen. Participants whose cultures included both a Gram-positive and a Gram-negative pathogen are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 62 | 8
percentage of participants
  Clinical Cure | 96.8 [88.8 to 99.6] | 87.5 [47.3 to 99.7]
  Clinical Failure | 0.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 12.5 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.
  Indeterminate | 3.2 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 0.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.

6. Secondary Outcome: Percentage of Participant With Clinical Response at Day 180 in the mITT Population
Description: as for outcome 1
Time Frame: Day 180
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 67 | 8
percentage of participants
  Clinical Cure | 94.0 [85.4 to 98.3] | 87.5 [47.3 to 99.7]
  Clinical Failure | 3.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 0.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.
  Indeterminate | 3.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 12.5 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.

7. Secondary Outcome: Percentage of Participants With Clinical Response at Day 180 in the CE Population
Description: as for outcome 1
Time Frame: Day 180
Population: CE-D180 population included all mITT participants who met specific conditions for evaluability at Day 180 (D180).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 66 | 8
percentage of participants
  Clinical Cure | 95.5 [87.3 to 99.1] | 87.5 [47.3 to 99.7]
  Clinical Failure | 1.5 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 0.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.
  Indeterminate | 3.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 12.5 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.

8. Secondary Outcome: Percentage of Participants With Clinical Response at Day 365 in the mITT Population
Description: as for outcome 1
Time Frame: Day 365
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 67 | 8
percentage of participants
  Clinical Cure | 94.0 [85.4 to 98.3] | 87.5 [47.3 to 99.7]
  Clinical Failure | 3.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.
  Indeterminate | 3.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 12.5 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.

9. Primary Outcome: Percentage of Participants With Clinical Response at Day 365 in the CE Population
Description: as for outcome 1
Time Frame: Day 365
Population: CE-D365 population included all mITT participants who met specific conditions for evaluability at Day 365 (D365).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 66 | 8
percentage of participants
  Clinical Cure | 95.5 [87.3 to 99.1] | 87.5 [47.3 to 99.7]
  Clinical Failure | 1.5 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.
  Indeterminate | 3.0 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure. | 12.5 [NA to NA] — As per protocol, 95% CI was only calculated for outcome of clinical cure.

10. Secondary Outcome: Number of Participants With Clinical Cure by Baseline Pathogen at Day 42 in the CE Population
Description: as for outcome 1
Time Frame: Day 42
Population: CE-D42 population included all mITT participants who met specific conditions for evaluability at Day 42 (D42). Includes participants who had baseline pathogens. Participants who had more than one pathogen at Baseline were counted in each category.
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 62 | 8
participants
  Staphylococcus aureus: number analyzed (Participants) | 42 | 6
  Staphylococcus aureus | 41 | 5
  Staphylococcus epidermidis: number analyzed (Participants) | 6 | 2
  Staphylococcus epidermidis | 6 | 2
  Staphylococcus haemolyticus: number analyzed (Participants) | 4 | 0
  Staphylococcus haemolyticus | 3 |
  Staphylococcus pasteuri: number analyzed (Participants) | 1 | 0
  Staphylococcus pasteuri | 1 |
  Staphylococcus hominis: number analyzed (Participants) | 2 | 0
  Staphylococcus hominis | 1 |
  Staphylococcus simulans: number analyzed (Participants) | 1 | 0
  Staphylococcus simulans | 1 |
  Enterococcus faecalis: number analyzed (Participants) | 7 | 1
  Enterococcus faecalis | 7 | 1
  Enterococcus faecium: number analyzed (Participants) | 1 | 0
  Enterococcus faecium | 1 |
  Streptococcus agalactiae: number analyzed (Participants) | 1 | 1
  Streptococcus agalactiae | 1 | 1
  Streptococcus dysgalactiae: number analyzed (Participants) | 1 | 0
  Streptococcus dysgalactiae | 1 |
  Streptococcus pyogenes: number analyzed (Participants) | 1 | 0
  Streptococcus pyogenes | 1 |
  Corynebacterium striatum: number analyzed (Participants) | 2 | 1
  Corynebacterium striatum | 2 | 1
  Aerococcus viridans: number analyzed (Participants) | 1 | 0
  Aerococcus viridans | 1 |
  Globicatella species: number analyzed (Participants) | 1 | 0
  Globicatella species | 1 |
  Micrococcus luteus: number analyzed (Participants) | 1 | 0
  Micrococcus luteus | 1 |
  Peptoniphilus harei: number analyzed (Participants) | 2 | 0
  Peptoniphilus harei | 2 |
  Anaerococcus prevotii: number analyzed (Participants) | 1 | 0
  Anaerococcus prevotii | 1 |
  Finegoldia magna: number analyzed (Participants) | 1 | 0
  Finegoldia magna | 1 |
  Peptostrep. anaerobius: number analyzed (Participants) | 1 | 0
  Peptostrep. anaerobius | 1 |
  Escherichia coli: number analyzed (Participants) | 3 | 0
  Escherichia coli | 3 |
  Klebsiella pneumoniae: number analyzed (Participants) | 2 | 1
  Klebsiella pneumoniae | 2 | 1
  Pseudomonas aeruginosa: number analyzed (Participants) | 2 | 1
  Pseudomonas aeruginosa | 2 | 0
  Enterobacter cloacae complex: number analyzed (Participants) | 2 | 0
  Enterobacter cloacae complex | 2 |
  Morganella morganii: number analyzed (Participants) | 2 | 0
  Morganella morganii | 2 |
  Proteus mirabilis: number analyzed (Participants) | 1 | 1
  Proteus mirabilis | 1 | 1
  Raoultella planticola: number analyzed (Participants) | 1 | 1
  Raoultella planticola | 1 | 0
  Serratia marcescens: number analyzed (Participants) | 0 | 1
  Serratia marcescens |  | 0
  Escherichia hermannii: number analyzed (Participants) | 1 | 0
  Escherichia hermannii | 1 |
  Pluralibacter gergoviae: number analyzed (Participants) | 1 | 0
  Pluralibacter gergoviae | 1 |
  Acinetobacter calcoaceticus: number analyzed (Participants) | 1 | 0
  Acinetobacter calcoaceticus | 1 |
  Bacteroides fragilis: number analyzed (Participants) | 2 | 0
  Bacteroides fragilis | 2 |
  Bacteroides thetaiotaomicron: number analyzed (Participants) | 1 | 0
  Bacteroides thetaiotaomicron | 1 |
  Bacteroides vulgatus: number analyzed (Participants) | 1 | 0
  Bacteroides vulgatus | 1 |
  Porphyromonas asaccharolytica: number analyzed (Participants) | 2 | 0
  Porphyromonas asaccharolytica | 2 |
  Prevotella melaninogenica: number analyzed (Participants) | 2 | 0
  Prevotella melaninogenica | 2 |
  Prevotella disiens: number analyzed (Participants) | 1 | 0
  Prevotella disiens | 1 |
  Prevotella intermedia: number analyzed (Participants) | 1 | 0
  Prevotella intermedia | 1 |
  Prevotella species: number analyzed (Participants) | 1 | 0
  Prevotella species | 1 |

11. Secondary Outcome: Number of Participants With Clinical Cure by Baseline Pathogen at Day 180 in the CE Population
Description: as for outcome 1
Time Frame: Day 180
Population: CE-D180 population included all mITT participants who met specific conditions for evaluability at Day 180 (D180). Includes participants who had baseline pathogens. Participants who had more than one pathogen at Baseline were counted in each category.
Measure: Number; unit: participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 61 | 8
participants
  Staphylococcus aureus: number analyzed (Participants) | 41 | 6
  Staphylococcus aureus | 39 | 5
  Staphylococcus epidermidis: number analyzed (Participants) | 6 | 2
  Staphylococcus epidermidis | 6 | 2
  Staphylococcus haemolyticus: number analyzed (Participants) | 4 | 0
  Staphylococcus haemolyticus | 3 |
  Staphylococcus pasteuri: number analyzed (Participants) | 1 | 0
  Staphylococcus pasteuri | 1 |
  Staphylococcus hominis: number analyzed (Participants) | 2 | 0
  Staphylococcus hominis | 1 |
  Staphylococcus simulans: number analyzed (Participants) | 1 | 0
  Staphylococcus simulans | 1 |
  Enterococcus faecalis: number analyzed (Participants) | 7 | 1
  Enterococcus faecalis | 7 | 0
  Enterococcus faecium: number analyzed (Participants) | 1 | 0
  Enterococcus faecium | 1 |
  Streptococcus agalactiae: number analyzed (Participants) | 1 | 1
  Streptococcus agalactiae | 1 | 1
  Streptococcus dysgalactiae: number analyzed (Participants) | 1 | 0
  Streptococcus dysgalactiae | 1 |
  Streptococcus pyogenes: number analyzed (Participants) | 1 | 0
  Streptococcus pyogenes | 1 |
  Corynebacterium striatum: number analyzed (Participants) | 2 | 1
  Corynebacterium striatum | 2 | 1
  Aerococcus viridans: number analyzed (Participants) | 1 | 0
  Aerococcus viridans | 1 |
  Globicatella species: number analyzed (Participants) | 1 | 0
  Globicatella species | 1 |
  Micrococcus luteus: number analyzed (Participants) | 1 | 0
  Micrococcus luteus | 1 |
  Peptoniphilus harei: number analyzed (Participants) | 2 | 0
  Peptoniphilus harei | 2 |
  Anaerococcus prevotii: number analyzed (Participants) | 1 | 0
  Anaerococcus prevotii | 1 |
  Finegoldia magna: number analyzed (Participants) | 1 | 0
  Finegoldia magna | 1 |
  Peptostrep. anaerobius: number analyzed (Participants) | 1 | 0
  Peptostrep. anaerobius | 1 |
  Escherichia coli: number analyzed (Participants) | 3 | 0
  Escherichia coli | 3 |
  Klebsiella pneumoniae: number analyzed (Participants) | 2 | 1
  Klebsiella pneumoniae | 2 | 1
  Pseudomonas aeruginosa: number analyzed (Participants) | 2 | 1
  Pseudomonas aeruginosa | 2 | 1
  Enterobacter cloacae complex: number analyzed (Participants) | 2 | 0
  Enterobacter cloacae complex | 2 |
  Morganella morganii: number analyzed (Participants) | 2 | 0
  Morganella morganii | 2 |
  Proteus mirabilis: number analyzed (Participants) | 1 | 1
  Proteus mirabilis | 1 | 1
  Raoultella planticola: number analyzed (Participants) | 1 | 1
  Raoultella planticola | 1 | 1
  Serratia marcescens: number analyzed (Participants) | 0 | 1
  Serratia marcescens |  | 1
  Escherichia hermannii: number analyzed (Participants) | 1 | 0
  Escherichia hermannii | 1 |
  Pluralibacter gergoviae: number analyzed (Participants) | 1 | 0
  Pluralibacter gergoviae | 1 |
  Acinetobacter calcoaceticus: number analyzed (Participants) | 1 | 0
  Acinetobacter calcoaceticus | 1 |
  Bacteroides fragilis: number analyzed (Participants) | 2 | 0
  Bacteroides fragilis | 2 |
  Bacteroides thetaiotaomicron: number analyzed (Participants) | 1 | 0
  Bacteroides thetaiotaomicron | 1 |
  Bacteroides vulgatus: number analyzed (Participants) | 1 | 0
  Bacteroides vulgatus | 1 |
  Porphyromonas asaccharolytica: number analyzed (Participants) | 2 | 0
  Porphyromonas asaccharolytica | 2 |
  Prevotella melaninogenica: number analyzed (Participants) | 2 | 0
  Prevotella melaninogenica | 2 |
  Prevotella disiens: number analyzed (Participants) | 1 | 0
  Prevotella disiens | 1 |
  Prevotella intermedia: number analyzed (Participants) | 1 | 0
  Prevotella intermedia | 1 |
  Prevotella species: number analyzed (Participants) | 1 | 0
  Prevotella species | 1 |

ADVERSE EVENTS:
Time Frame: From Baseline (Day 0) to Day 365
Arm/Group | Dalbavancin | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/70 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/70 | 0/10
Other Adverse Events (participants affected / at risk) | 0/70 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalbavancin (N=70) | Standard of Care (N=10)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that the first results publication shall be made in conjunction with a joint multi-center publication. If the multi-center publication is not submitted within 12 months after conclusion of the study at all sites, or if the sponsor confirms not to publish the results, the PI may publish the results from the institution subject to terms of the clinical trial agreement. The publication must be sent to Sponsor at least 60 days before the intended submission date for reference and comment.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT02685033/SAP_000.pdf
  • Study Protocol (2015-06-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT02685033/Prot_001.pdf